CLINICAL TRIAL: NCT04482387
Title: DigiVis: Validation of Self-testing Visual Acuity Web-based App to Aid Ophthalmic Telephone Consultations During Covid19 Lockdown and Subsequent Social Distancing Crisis
Brief Title: DigiVis: Self-testing Vision App for Telephone Consultations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Louise Allen, Principal investigator, Cambridge University Hospitals NHS Foundation Trust
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: IRAS196573
Record Dates: First submitted 2020-07-17; First posted 2020-07-22 (Actual); Results first posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-02

CONDITIONS: Visual Impairment; Amblyopia Suspect
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Intervention Model Description: Patients will test their own vision twice using the DigiVis app twice, subsequently they will have visual acuity assessment in eye clinic by a trained examiner. The results of visual acuity will be compared using Bland Altman statistical analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects recruited to visual acuity testing (Other): All recruited subjects will have the intervention (Digivis visual acuity self-testing) and the standard clinical visual acuity assessment in clinic.
  Interventions: Device: DigiVis visual acuity app

INTERVENTIONS:
Device: DigiVis visual acuity app — Self-testing of visual acuity app on two occasions

SUMMARY:
This trial aims to assess the accuracy and test-retest variability of a new digital app which enables community visual acuity testing without requirement of an trained examiner.

DETAILED DESCRIPTION:
Eye problems like macular degeneration and amblyopia (lazy eye) require regular monitoring to prevent permanent visual impairment. Over 2000 patients a month are seen in Cambridge University Hospitals National Health Service Trust (CUH) eye clinics; concern about Covid-19 infection has led to over 80% of consultations being conducted by telephone with few clinical clues to inform decision making. Patients will face long delays even when routine clinics restart: there is no doubt that some will suffer preventable visual loss.

DigiVis is a web-based vision testing app enabling self-testing of vision at home. Early testing and patient feedback is positive: 80% of children prefer DigiVis to regular testing. The investigators wish to test how accurately the app works for home use, by asking older children and adults to self-test their vision prior to their planned face to face clinic appointment. Once tested, DigiVis will be available free of charge to patients, not only during the Covid-19 crisis, but also to support telephonic consultations in the future.

Visual acuity (VA) is a fundamental measure of vision required for all ophthalmic assessments. It is measured by health professionals using vision charts. DigiVis is a new app which enables self-testing of VA using two wirelessly connected digital devices. By matching letters on a handheld device to those displayed on the second device a distance away, threshold VA can be measured using a staircase algorithm. The distance and scaling of the test is vital to its accuracy and a concept (patent filed by Cambridge Enterprise) in DigiVis enables this without the need for manual distance measurement or an observer.

Early validation using two tablet computers in 150 clinic patients has given positive results, both in testing accuracy and patient feedback. With the current Covid-19 crisis limiting face to face appointments, there is an urgent need for accurate home VA assessment. The DigiVis app has been re-coded for free website delivery for this purpose.

The investigators wish to formally validate DigiVis home testing following Conformitè Europëenne (CE class I) marking so that it can be recommended for clinical use. 250 patients will be invited to self-test their VA twice using DigiVis prior to a planned face to face clinic appointment. The test-retest variability and comparison of DigiVis VA to chart based assessment will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Age between 5 and 85 years
* Previous recorded visual acuity of at least +0.8 logMAR in or both eyes

Exclusion Criteria:

* Individuals with poor conversant English
* Individuals with cognitive impairment
* Subjects unable to access the internet on two digital devices

Ages: 5 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen E Kelleher, Study Director — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Cambridge University Hospitals NHS Trust, Cambridge, Cambs, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rono HK, Bastawrous A, Macleod D, Wanjala E, Di Tanna GL, Weiss HA, Burton MJ. Smartphone-based screening for visual impairment in Kenyan school children: a cluster randomised controlled trial. Lancet Glob Health. 2018 Aug;6(8):e924-e932. doi: 10.1016/S2214-109X(18)30244-4. PMID 30012273
- [Background] Bastawrous A, Rono HK, Livingstone IA, Weiss HA, Jordan S, Kuper H, Burton MJ. Development and Validation of a Smartphone-Based Visual Acuity Test (Peek Acuity) for Clinical Practice and Community-Based Fieldwork. JAMA Ophthalmol. 2015 Aug;133(8):930-7. doi: 10.1001/jamaophthalmol.2015.1468. PMID 26022921
- [Background] Thirunavukarasu AJ, Mullinger D, Rufus-Toye RM, Farrell S, Allen LE. Clinical validation of a novel web-application for remote assessment of distance visual acuity. Eye (Lond). 2022 Oct;36(10):2057-2061. doi: 10.1038/s41433-021-01760-2. Epub 2021 Aug 30. PMID 34462579

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Over a two month period, research administrators posted study invitations and information leaflets to all patients due to attend an eye clinic appointment. Inclusion criteria were: age over 4 years, VA of +0.8 (6/38 Snellen) or better in each eye and no documentation of cognitive disability. The clinician researcher phoned the patient to explain the study, take verbal consent and give password access to the DigiVis test.
Pre-assignment Details: All participants underwent both the DigiVis testing and the standard clinical visual acuity test.
Units Other Than Participants: Eyes
Groups:
- All Study Participants: Right eye data for all 120 participants to the study.
Period: Overall Study
Arm/Group | All Study Participants
Started | 120; 120 Eyes
Completed | 120; 120 Eyes
Not Completed | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 120
Age, Customized [Count of Participants; unit: Participants]
  Age category: 5-10 years | 44
  Age category: 11-54 years | 37
  Age category: 55 - 75 years | 32
  Age category: 76-85 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 54
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Mean Bias Between the Difference Between DigiVis and Standard Visual Assessment Compared to the Mean of DigiVis and Standard Visual Assessment
Description: The mean bias (difference) in visual acuity assessment score between the difference in DigiVis and standard testing in logMAR units and the mean of DigiVis and standard testing in logMAR units was calculated. Where 0.00 logMAR is the value representing perfect distance visual acuity (equivalent to 20/20 Snellen acuity) and 1.00 logMAR is the value representing worst distance visual acuity (equivalent to 20/200 Snellen acuity).
Time Frame: within 30 days
Population: All participants had their right eye tested firstly with the standard chart technique and subsequently with DigiVis
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- Standard Vision Testing: Participants had standard chart testing of their right eye.
- DigiVis Vision Testing: The same cohort of patients then had DigiVis vision testing
Arm/Group | Standard Vision Testing | DigiVis Vision Testing
Number analyzed (Participants) | 120 | 120
logMAR | 0.112 (0.247) | 0.100 (0.270)

2. Secondary Outcome: Mean Bias Between Repeated DigiVis Test Assessments
Description: Mean bias between the difference of two DigiVis visual acuity assessments compared to the mean of two digiVis assessments measured in logMAR units.
Time Frame: within 30 days
Population: Participants able to undertake DigiVis testing twice to analyse test repeatability
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- First DigiVis Test: Patients undertaking DigiVis testing for the first time
- Repeated DigiVis Testing: Patients undertaking DigiVis a second time
Arm/Group | First DigiVis Test | Repeated DigiVis Testing
Number analyzed (Participants) | 105 | 105
logMAR | 0.100 (0.270) | 0.105 (0.258)

ADVERSE EVENTS:
Time Frame: uo to 60 days
Description: No adverse events
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/120
Serious Adverse Events (participants affected / at risk) | 0/120
Other Adverse Events (participants affected / at risk) | 0/120

LIMITATIONS AND CAVEATS:
The study recruited a smaller number of participants than originally intended but 120 participants was sufficient to enable narrow 95% confidence limits.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-15): https://cdn.clinicaltrials.gov/large-docs/87/NCT04482387/Prot_SAP_000.pdf